CLINICAL TRIAL: NCT00641030
Title: A Phase I Study of Clofarabine Plus High Dose Melphalan as a Conditioning Regimen for Allogeneic Transplantation
Brief Title: Clofarabine and High-Dose Melphalan Followed by Donor Stem Cell Transplant in Patients With Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06114; P30CA033572 (NIH); CHNMC-06114; CDR0000589304 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-03-20; First posted 2008-03-21 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; childhood myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine; Melphalan; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clofarabine — Administered at the appropriate dose level(dose level one = 30 mg/m2, dose level two and three = 40 mg/m2)on days -9 to day -5 from transplant
Drug: melphalan — Administered at the appropriate dose level (dose level one and two = 100 mg/m2, dose level three = 140 mg/m2) on day -4 from transplant
Genetic: gene expression analysis — Peripheral blood draw on day -9 and day -4 prior to transplant
Genetic: reverse transcriptase-polymerase chain reaction — Peripheral blood draw on day -9 and day -4 prior to transplant
Other: flow cytometry — Bone marrow aspirate and biopsy to confirm diagnosis prior to transplant, day -9 pre-transplant, day 30 post-transplant, day 100 post-transplant, 6 months post-transplant, one year post-transplant, then yearly through year 5 post-transplant
Other: laboratory biomarker analysis — Peripheral blood draw day -9 or earlier pre-transplant, day 14 post-transplant, day 30 post-transplant, day 60 post-transplant, day 100 post-transplant, 6 months and one year post-transplant.
Procedure: allogeneic hematopoietic stem cell transplantation — Infusion of allogeneic hematopoietic stem cells on day 0 of transplant

SUMMARY:
RATIONALE: Giving chemotherapy, such as clofarabine and melphalan, before a donor stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine when given together with high-dose melphalan followed by a donor stem cell transplant in treating patients with acute myeloid leukemia, acute lymphocytic leukemia, or myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose and toxicities of clofarabine when administered with high-dose melphalan as a conditioning regimen in patients undergoing allogeneic stem cell transplantation for acute myeloid leukemia, acute lymphocytic leukemia, or myelodysplastic syndromes.
* To assess the efficacy of this regimen in facilitating engraftment in these patients.
* To perform correlative laboratory studies of engraftment, immune reconstitution, and therapeutic outcomes.

OUTLINE: This is a dose-escalation study of clofarabine. Patients are stratified according to age (< 18 years vs ≥ 18 years).

* Reduced-intensity conditioning regimen: Patients receive clofarabine IV over 30 minutes on days -9 to -5 and high-dose melphalan IV over 30 minutes on day -4.

Cohorts of 3-6 patients receive escalating doses of clofarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Allogeneic stem cell transplantation: Patients undergo allogeneic stem cell transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 10 hours or orally twice daily beginning on day -1 and continuing until day 90-100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV or orally twice daily beginning on day 0 and continuing until day 28, followed by a taper in the absence of GVHD.

Patients undergo blood and/or bone marrow sample collection periodically for correlative laboratory studies. Samples are examined for markers of immune reconstitution (i.e., CD8+ T lymphocytes, CD4+ T lymphocytes, NK cells, B cells, and monocytes) by flow cytometry and for diversity of the reconstituted T-cell repertoire by PCR-based T-cell receptor repertoire analysis. Samples are also examined for gene expression of hRRM2 and markers of apoptosis (i.e., Bcl-2, Bid, NFkB2, and Bcl-3) by real-time RT-PCR and for markers of ribonucleotide reductase inhibition (i.e., dCTP levels in circulating peripheral blood mononuclear cells).

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Acute myeloid leukemia
  * Acute lymphocytic leukemia
  * Myelodysplastic syndromes
* Disease meets 1 of the following criteria:

  * In first complete remission (CR)
  * In second CR
  * In relapse
* No more than 50% blasts in bone marrow
* Not deemed eligible for standard transplantation regimens by the attending physician, or at high risk for relapse
* No suspected or proven CNS leukemia
* HLA-matched (6/6) sibling donor available

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Glomerular filtration rate (pediatric patients) or creatinine clearance ≥ 60 mL/min OR serum creatinine < 1.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times ULN
* LVEF ≥ 50% by ECHO or MUGA scan
* DLCO or FEV_1 ≥ 40% predicted
* Not pregnant
* Negative pregnancy test
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing, active, or poorly controlled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Poorly controlled pulmonary disease
  * Psychiatric illness/social situation that would limit compliance with study requirement
* No active cytomegalovirus (CMV) or fungal disease
* HIV negative

PRIOR CONCURRENT THERAPY:

* Recovered from prior intensive chemotherapy (pediatric patients)
* At least 100 days since prior autologous stem cell transplantation
* At least 100 days since prior radiotherapy administered as part of a transplantation conditioning regimen
* At least 4 weeks since prior chemotherapy
* At least 24 hours since prior hydroxyurea for blast count control

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 weeks from the start of treatment
Dose-limiting toxicity as assessed by NCI CTCAE v3.0 and the Modified Bearman scale | 4 weeks from the start of treatment
Graft failure or rejection | 35 days post-transplant

SECONDARY OUTCOMES:
Efficacy | One year post-transplant
Correlative laboratory studies of engraftment, immune reconstitution, and therapeutic outcomes | One year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Stein, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States